CLINICAL TRIAL: NCT01220427
Title: Micro-RNA Expression Profiles in High Risk Prostate Cancer
Status: Terminated | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Martin Spahn, University Hospital Würzburg
Other Study IDs: mi-RNA HR-Pca
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2010-08

CONDITIONS: Prostate Cancer; Radical Prostatectomy
Keywords: high-risk prostate cancer; radical prostatectomy; micro-RNA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical high-risk prostate cancer, radical prostatectomy

SUMMARY:
The purpose of this study is to determine whether specific Micro-RNA expression profiles are related to Prostate cancer outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically localised high risk prostate cancer (cT>2, bx GS >7, PSA >20 ng/ml) scheduled for radical prostatectomy.

Exclusion Criteria:

Non high risk prostate cancer

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospital, community hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Recurrence free survival | Yearly update until clinical progression
  The patients will be followed in regular time intervals in accordance with the EAU-Guidelines (2010) and the S-3 Guideline for Prostate cancer of the German Urological Association. Data will be updated once yearly for until death.

SECONDARY OUTCOMES:
Cancer specific survival | Yearly update until death
  The patients will be followed in regular time intervals in accordance with the EAU-Guidelines (2010) and the S-3 Guideline for Prostate cancer of the German Urological Association. Data will be updated once yearly until death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Pediatric Urology University Hospital Würzburg, Würzburg, Germany